CLINICAL TRIAL: NCT03007316
Title: Clinical Evaluation of Soft Tissue Esthetics Around Immediate Implants in Vascularized Interpositional Periosteal Connective Tissue Grafted Versus Non-grafted Sites. A Randomized Controlled Clinical Trial.
Brief Title: Evaluation of Esthetics Around Immediate Implants in VIP - CT Grafted vs Non-grafted Sites.RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzy Nabil Naiem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0
Record Dates: First submitted 2016-12-23; First posted 2017-01-02 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Buccal Bone Loss in Immediate Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Implants + VIP graft. (Experimental): Immediate implants placed with simultaneous vascularized interpositional periosteal (VIP) connective tissue graft augmentation.
  Interventions: Procedure: VIP graft
- Immediate Implants only (No Intervention): Immediate Implants only without soft tissue augmentation.

INTERVENTIONS:
Procedure: VIP graft — surgical soft tissue grafting concomitant to implant placement
  Arms: Immediate Implants + VIP graft.

SUMMARY:
An array of soft tissue augmentation techniques have been employed concomitant to implant placement, as free connective tissue grafts or pedicle grafts for keratinized tissue thickening in attempt not only to augment the soft tissue for better resistance to inflammation and improved esthetic stability, but to preserve buccal bone thickness as well.

Results obtained from the literature were controversial regarding the need of soft tissue augmentation to curb buccal bone resorption and preserve pink esthetics. Scarce literature was found, that monitored the ridge alterations following implant placement.

Our study will monitor the effect of soft tissue augmentation on soft tissue esthetics and buccal bone resorption during the process of remodeling in a measurable way.

DETAILED DESCRIPTION:
Alveolar bone remodeling following extraction could not be prevented by immediate implant placement. Soft tissue augmentaion techniques have been suggested in order to overcome the alterations of buccal bone during remodeling. Nevertheless, it is still inconclusive whether soft tissue augmentation procedures actually have a protective role in preserving buccal bone thickness in immediate implants.

Aim is to clinically and radiographically assess the effect of soft tissue grafting on buccal bone resorption and pink esthetics around immediately placed implants in maxillary anterior teeth after 24 months following implant placement. 18 non-restorable maxillary anterior teeth randomly assigned into 2 groups: (test group) immediately placed implants with simultaneous vascular interpositional periosteal connective tissue (VIP-CT) grafting versus non-augmented implant sites (control group). Buccal bone changes were assessed at implant placement (0) and at 4,9,12 and 24 months from baseline by specially manufactured device and at 24 months by cone beam computed tomography scans (CBCT). Pink esthetic score (PES) was evaluated at 6, 9, 12 and 24 months intervals. Pain and satisfaction were assessed through questionnaires to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have at least one unrestorable tooth in the esthetic zone that needs to be extracted.
* Patients with healthy systemic condition.
* Buccal bone thickness should be at least 1mm.
* Availability of bone apical and palatal to the socket to provide primary stability.
* Good oral hygiene.

Exclusion Criteria:

* Patients with signs of acute infection related to the area of interest.
* Current and former smokers
* Pregnant.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
"PES" Pink Esthetic Score | 2 years
  esthetic assessment by the pink esthetic score introduced by furhauser et al 2005

CONTACTS AND LOCATIONS:
Overall Officials: Hani El Nahass, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Greater Cairo, Egypt